CLINICAL TRIAL: NCT04307654
Title: Evaluation of the Relationship Between Lactacidemia and Postoperative Complications After Cytoreduction Surgery for Peritoneal Carcinomatosis
Brief Title: Lactate and Complications in Cytoreduction Surgery for Peritoneal Carcinomatosis
Status: Completed | Type: Observational
Sponsor: Hospital General Universitario de Castellón (Other)
Responsible Party: Principal Investigator, Marta Soriano Hervás, Principal investigator, Hospital General Universitario de Castellón
Other Study IDs: HGCLAC01
Record Dates: First submitted 2020-03-09; First posted 2020-03-13 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Lactacidemia and Complications
Keywords: lactic acid; Cytoreductive surgery; postoperative complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Serum lactate is a risk factor for postoperative complications in patients undergoing cytoreduction surgery in peritoneal carcinomatosis

DETAILED DESCRIPTION:
Background. Cytoreduction surgery has been developed as a treatment of peritoneal carcinomatosis. However, this surgery is associated with important complications. The present study attempts to assess the relationship between lactacidemia levels and the rate of associated complications in patients undergoing cytoreduction surgery during the immediate postoperative period in a critical unit.

Methods. Retrospective observational study. 57 patients underwent cytoreduction surgery during the years 2014 and 2015 at the General University Hospital of Castellón. All patients were admitted to the critical unit immediately after surgery. Lactacidemia levels at the time of admission and discharge from the critical unit were collected. Post-surgical complications that appeared during the stay in the critical unit were recorded and classified according to the Clavien-Dindo classification.

Lactacidemia levels were still significantly higher in this group at the time of discharge.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with peritoneal carcinomatosis who underwent cytoreduction surgery in the Multidisciplinary Unit of Abdomino-Pelvic Oncology Surgery (MUAPOS) of the University General Hospital of Castellón.

Exclusion Criteria:

* patients without lactic acid levels in the register.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients diagnosed with peritoneal carcinomatosis who underwent cytoreduction surgery in the Multidisciplinary Unit of Abdomino-Pelvic Oncology Surgery (MUAPOS) of the University General Hospital of Castellón
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2014-06 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Postoperative complications | 2014-2016
  complications in patients undergoing cytoreduction surgery during the immediate postoperative period in the Intensive Care Unit (ICU) at the General Hospital of Castellón (HGCS) between 2014 and 2016.